CLINICAL TRIAL: NCT01572636
Title: MT2011-21C Laronidase (Aldurazyme TM) Enzyme Replacement Therapy (ERT) With Hematopoietic Stem Cell Transplantation (HSCT) for Hurler Syndrome (MPS IH).
Brief Title: Laronidase (Aldurazyme TM) Enzyme Replacement Therapy With Hematopoietic Stem Cell Transplant for Hurler Syndrome
Status: Terminated | Type: Observational
Why Stopped: Research Cancelled
Sponsor: Masonic Cancer Center, University of Minnesota (Other)
Responsible Party: Sponsor
Other Study IDs: 2011OC140; MT2011-21C (Other: Blood and Marrow Transplant Program)
Record Dates: First submitted 2012-04-04; First posted 2012-04-06 (Estimated); Last update posted 2018-09-27 (Actual); Status verified 2018-09

CONDITIONS: Mucopolysaccharidosis Type IH; MPS I; Hurler Syndrome
Keywords: Hurler Syndrome
MeSH Terms: conditions — Mucopolysaccharidosis I | interventions — Iduronidase

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Laronidase use in Hurler Syndrome: Laronidase receiving prior and post transplant
  Interventions: Drug: Laronidase

INTERVENTIONS:
Drug: Laronidase — Administered 0.58 mg/kg/dose intravenously (IV) once a week beginning 12 weeks before planned hematopoietic stem cell transplant (HSCT) and resume same dosing regimen for 8 weeks after HSCT.
  Other Names: Aldurazyme

SUMMARY:
This is a standard of care treatment guideline for patients with the diagnosis of mucopolysaccharidosis type IH (MPS I, Hurler syndrome) who are being considered as candidates for first hematopoietic stem cell transplantation (HSCT) according to a University of Minnesota myeloablative HSCT protocol.

DETAILED DESCRIPTION:
Laronidase Enzyme Replacement Therapy will be performed using laronidase once a week for 12 weeks prior to hematopoietic stem cell transplantation and for 8 weeks post-transplant to reduce pulmonary complications.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of mucopolysaccharidosis type IH (MPS I, Hurler syndrome) and being considered as a candidate for first transplant according to a University of Minnesota myeloablative hematopoietic stem cell transplant (HSCT) protocol

Exclusion Criteria:

* No prior therapy with laronidase enzyme replacement therapy (ERT)

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Diagnosis of mucopolysaccharidosis type IH (MPS I, Hurler syndrome) and being considered as a candidate for first transplant according to a University of Minnesota myeloablative hematopoietic stem cell transplant (HSCT) protocol
Sampling Method: Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2012-03-28 (Actual); Primary Completion 2018-05-01 (Actual); Study Completion 2018-05-01 (Actual)

PRIMARY OUTCOMES:
Overall Survival | At 1 Year
  Patients alive at 1 year post transplantation.

SECONDARY OUTCOMES:
Incidence of Engraftment | 1 Year Post Transplant
  The incidence of donor engraftment will be estimated by taking the simple proportion of patients achieving donor engraftment over the number of evaluable patients. Donor engraftment will be defined as achieving an absolute neutrophil count ≥ 5x10^8/kg for three consecutive days before day 42 and maintenance of >10% donor chimerism through one year post transplant or death.
Incidence of Grade III-IV Acute Graft Versus Host Disease | Day 100
  Cumulative incidence will be used to estimate grade III-IV acute GvHD, treating death as a competing risk.
Proportion of patients in need of ventilator support | 1 Year
  Count of patients using ventilator by 1 year.

CONTACTS AND LOCATIONS:
Overall Officials: Paul Orchard, M.D., Principal Investigator — Masonic Cancer Center, University of Minnesota
Locations (1):
- Masonic Cancer Center, University of Minnesota, Minneapolis, Minnesota, United States